CLINICAL TRIAL: NCT03309579
Title: Aneurysmal Subarachnoid Hemorrhage - Red Blood Cell Transfusion and Outcome (SAHaRA): A Randomized Controlled Trial
Brief Title: SAHaRA: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTO:903
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Aneurysmal subarachnoid hemorrhage (aSAH); Red Blood Cell Transfusion (RBC); Vasospasm; Intracranial Hemorrhages; Cardiovascular Diseases
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Hemorrhages; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Multicentre pragmatic, open-label blinded-endpoint
Who Masked: Outcomes Assessor
Masking Description: open-label blinded-endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal RBC Transfusion Strategy (Experimental): Hemoglobin value of ≤100g/L
  Interventions: Other: Liberal RBC Transfusion Strategy
- Restrictive RBC Transfusion Strategy (Active Comparator): Hemoglobin value of ≤80g/L
  Interventions: Other: Restrictive RBC Transfusion Strategy

INTERVENTIONS:
Other: Liberal RBC Transfusion Strategy — RBC transfusion is triggered by a Hemoglobin value of ≤100g/L
  Arms: Liberal RBC Transfusion Strategy
Other: Restrictive RBC Transfusion Strategy — Optional RBC transfusion is triggered by a Hemoglobin value of ≤80g/L
  Arms: Restrictive RBC Transfusion Strategy

SUMMARY:
The SAHaRA trial will clarify the role of treating anemia with Red Blood Cell (RBC) transfusion in a unique and vulnerable patient population, and determine whether that impacts on functional outcomes and mortality. It will guide best practice standards and clarify the optimal RBC transfusion strategy in patients with aSAH.

DETAILED DESCRIPTION:
We hypothesize that in adult patients suffering from aSAH and anemia, a liberal RBC transfusion strategy as compared to a restrictive RBC transfusion strategy decreases the combined rate of death and severe disability at 12 months (using the modified Rankin Scale)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old at time of SAH
2. First ever episode of aneurysmal SAH
3. Diagnosis of aSAH as confirmed by treating physician (eg: neurosurgeon or neuro- interventionalist) and supported by blood in subarachnoid space (e.g. cranial imaging or cerebrospinal fluid positive for xanthochromia, surgical visualization) that is the result of a ruptured aneurysm (e.g. direct visualization, cranial imaging or catheter angiogram)
4. Hb ≤100g/L within 10 days following aSAH (defined by first day of hospital presentation)

Exclusion Criteria:

1. Physician and or family decision to withdraw/withhold active medical care at time of enrolment
2. Active bleeding with hemodynamic instability at time of enrolment
3. Patients with contraindication or known objection to blood transfusions
4. SAH due to mycotic aneurysm, infundibulum and vascular malformations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 12 months post
  The Modified Rankin Scale (mRS) is a functional outcome measure in stroke. The interview consists of five sections: Constant Care, Assistance to Attend to Bodily Needs/For Walking, Assistance to Look After Own Affairs, Usual Duties and Activities and Symptoms as a Result of Stroke.
  The scale is scored from 0 reporting no symptoms at all, to 5 reporting severe disability. Death is indicated by a score of 6.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | 12 months post
  The Functional Independence Measure (FIM) assesses the level of a patient's disability considering the amount of support needed to care for them.Items are scored on the basis of how much assistance is required for the individual to carry out activities of daily living.
  The FIM is comprised of 18 items, grouped into 2 subscales - motor and cognition.
  Each item is scored on a 7 point ordinal scale, ranging from 1 to 7. The 2 subscales are then added to give a total FIM score between 18 and 126. The higher the score, the more independent the patient is in performing activities of daily living.
EuroQOL Quality of Life Scale (EQ5D) | 12 months post
  The EQ-5D measures generic health status. There are 5 dimensions: Mobility, Self-care, Usual Activities, Pain/Discomfort and Anxiety/Depression which are answered by 5 Problem Levels: None, Slight, Moderate, Severe and Unable. The result is a 5 digit number, 11111 indicating no problem in any dimension to 55555 indicating unable to complete in all dimensions.
  Quality of life is also assessed on a visual analog scale reported from 0 being the worst imaginable health status to 100 as the best imaginable health status.
Red Blood Cell Transfusions | up to 21 days
  The total number of red blood cell transfusions received.
Daily Hemoglobin | up to 21 days
  The lowest daily hemoglobin values.
Transfusion-related Complications | up to 28 days
  Complications such as Acute Respiratory Distress Syndrome (ARDS), cardiovascular failure, cardiac ischemia, deep venous thrombosis, pulmonary embolism, sepsis, and septic shock.
Delayed Cerebral Ischemia and Vasospasm | up to 28 days
  The incidence and severity of delayed cerebral ischemia and vasospasm.
Cerebral Infarction | up to 28 days
  The incidence of cerebral infarctions.
Mechanical Ventilation | up to 21 days
  If required, the duration of mechanical ventilation.
Length of Stay | 12 months post
  The length of ICU or hospital stay.
Mortality | 12 months post
  The number of deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Shane English, MD MSc FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (23):
- United States (3):
  - University of Colorado School of Medicine, Aurora, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
- Australia (5):
  - Nepean Hospital, Kingswood, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - The Alfred, Melbourne, Victoria
- Canada (15):
  - Foothills Medical Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Winnipeg Health Sciences Center, Winnipeg, Manitoba
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences Center, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Center, London, Ontario
  - Shane English, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - Centre hospitalier universitaire de Québec-Université Laval, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] English SW, Delaney A, Fergusson DA, Chasse M, Turgeon AF, Lauzier F, Tuttle A, Sadan O, Griesdale DE, Redekop G, Chapman M, Hannouche M, Kramer A, Seppelt I, Udy A, Kutsogiannis DJ, Zarychanski R, D'Aragon F, Boyd JG, Salt G, Bellapart J, Wood G, Cava L, Pickett G, Koffman L, Watpool I, Bass F, Hammond N, Ramsay T, Mallick R, Scales DC, Andersen CR, Fitzgerald E, Talbot P, Dowlatshahi D, Sinclair J, Acker J, Marshall SC, McIntyre L; SAHARA Trial Investigators on behalf of the Canadian Critical Care Trials Group; Canadian Critical Care Trials Group. Liberal or Restrictive Transfusion Strategy in Aneurysmal Subarachnoid Hemorrhage. N Engl J Med. 2025 Mar 13;392(11):1079-1088. doi: 10.1056/NEJMoa2410962. Epub 2024 Dec 9. PMID 39655786
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836

DOCUMENTS (2):
  • Study Protocol (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT03309579/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT03309579/SAP_002.pdf